CLINICAL TRIAL: NCT05598905
Title: Combined Effect of Pregabalin and Oxycodone, and Lacosamide and Oxycodone, on Breathing: an Exploratory Study in Healthy Volunteers (The Polo Study)
Brief Title: Combined Effect of Pregabalin and Oxycodone, and Lacosamide and Oxycodone, on Breathing
Acronym: POLO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Albert Dahan, Professor, Leiden University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: P22.044
Record Dates: First submitted 2022-10-13; First posted 2022-10-28 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Opioid-induced Respiratory Depression
Keywords: Oxycodone; Pregabalin; Lacosamide
MeSH Terms: interventions — Pregabalin; Oxycodone; Lacosamide

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized cross-over design.
  Amendment:
  In order to get an impression of the effect of 10 mg oxycodone per se, one open label arm of just 10 mg oxycodone as a visit 3 was added.
Who Masked: Participant, Investigator
Masking Description: Double-blind cross-over trial in which the order of visits is randomized.
  Amendment:
  In order to get an impression of the effect of 10 mg oxycodone per se, one open label arm of just 10 mg oxycodone as a visit 3 was added.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxycodone + Pregabalin (Experimental): Participants will visit twice. On one visit they will take a 10mg oxycodone tablet and 90 minutes later a 150mg pregabaline capsule.
  Interventions: Drug: Pregabalin 150mg; Drug: Oxycodone 10mg
- Oxycodone + Lacosamide (Experimental): Participants will visit twice. On one visit they will take a 10mg oxycodone tablet and 90 minutes later a 150mg Lacosamide capsule.
  Interventions: Drug: Oxycodone 10mg; Drug: Lacosamide 150 mg
- Oxycodone (Other): Amendment:
  one open label arm.
  In order to get an impression of the effect of 10 mg oxycodone per se, one open label arm of just 10 mg oxycodone as a visit 3 was added.
  Interventions: Drug: Oxycodone 10mg

INTERVENTIONS:
Drug: Pregabalin 150mg — one capsule of 150mg 90 minutes after 10mg of oxycodone
  Other Names: Lyrica capsule 150 mg
  Arms: Oxycodone + Pregabalin
Drug: Oxycodone 10mg — one 10mg tablet
  Other Names: Oxycodone tablet 10 mg
Drug: Lacosamide 150 mg — one capsule of 150mg 90 minutes after 10mg of oxycodone
  Other Names: Vimpat 150 mg capsule
  Arms: Oxycodone + Lacosamide

SUMMARY:
Opioids are commonly prescribed for moderate to severe pain. While initially intended for moderate to severe acute and cancer pain, opioids are currently frequently considered and prescribed in chronic noncancer pain. Due to the large increase in opioid prescription rate, the number of unintentional drug overdoses is rapidly increasing, not only in the Unites States but also in the Netherlands. A potential lethal consequence of an opioid overdose is opioid-induced respiratory depression. Additionally, it is well known that opioids are often used (and abused) in combination with other legal or illicit substances, for example alcohol, benzodiazepines, cannabis, neuropathic pain medication including the anticonvulsant pregabaline. There are no high-quality data on the interaction between oxycodone and (neuropathic pain) medication on the ventilatory control system. Case reports and randomized studies show that pregabalin induces respiratory depression when combined with opioids. Some alternatives to pregabalin may have a better safety profile. One such alternative is lacosamide, an antiepileptic with a different mode of action than pregabalin, and effective in the treatment of neuropathic pain. The hypothesis is that in contrast to lacosamide, pregabalin will increase the respiratory depressant effect of low-dose oxycodone.

The objective of the study is to quantify the effect of pregabalin and lacosamide on oxycodone-induced respiratory depression.

24 participants will be screened beforehand if subjects meet the inclusion and exclusion criteria. If so, the subjects will visit the hospital twice. On both occasions, participants will take a 10 mg oxycodone tablet and 90 minutes after a capsule of pregabalin or lacosamide. The order of visits will be randomized. During the visits, at set time points the hypercapnic ventilatory response will be measured, relief of nociception, pupil diameter and several side effects other than respiratory depression. There will be a washout period of 7 days between study visits with the study ending after 2 visits.

Amendment:

In order to get an impression of the effect of 10 mg oxycodone per se, one open label arm of just 10 mg oxycodone was added as a visit 3. Since the procedures in this third arm will be identical to the two blinded arms, no changes will be made to any of the procedures apart from not administering any lacosamide or pregabalin.

DETAILED DESCRIPTION:
Opioids are commonly prescribed for moderate to severe pain. While initially intended for moderate to severe acute and cancer pain, opioids are currently frequently considered and prescribed in chronic noncancer pain. Due to the large increase in opioid prescription rate, the number of unintentional drug overdoses is rapidly increasing, not only in the Unites States but also in the Netherlands. A potential lethal consequence of an opioid overdose is opioid-induced respiratory depression. Additionally, it is well known that opioids are often used (and abused) in combination with other legal or illicit substances, for example alcohol, benzodiazepines, cannabis, neuropathic pain medication including the anticonvulsant pregabalin. There are no high-quality data on the interaction between oxycodone and (neuropathic pain) medication on the ventilatory control system. Case reports and randomized studies show that pregabalin induces respiratory depression when combined with opioids. Some alternatives to pregabalin may have a better safety profile. One such alternative is lacosamide, an antiepileptic with a different mode of action than pregabalin, and effective in the treatment of neuropathic pain. The hypothesis is that in contrast to lacosamide, pregabalin will increase the respiratory depressant effect of low-dose oxycodone.

The objective of the study is to quantify the effect of pregabalin and lacosamide on oxycodone-induced respiratory depression.

24 participants will be screened beforehand if the subject meets the inclusion and exclusion criteria. If so, the subjects will visit the hospital twice. On both occasions, participants will be sober and take a 10 mg oxycodone tablet and 90 minutes after a capsule of pregabalin or lacosamide. The order of visits will be randomized using a randomisation list made in R by an independent investigator not involved in data acquisition. Upon arrival in the laboratory, a urinary drug test and breath alcohol test will be performed. When these tests are positive, the subject is excluded from further participation. An intravenous access line will be placed in the left or right arm/hand for fluid administration (NaCl/Glucose 50-100 ml/h). Next, the first hypercapnic ventilatory responses (HCVR) will be obtained (t = -30 min). This is the pre-dug baseline measurement. At t = 0, the subjects will next receive a 10 mg oxycodone immediate release tablet that the subjects will swallow with 100 mL water. Next, the HCVRs at 1-hour intervals will be obtained until 8 hours after oxycodone intake. At t = 90 min the subject will ingest a pregabalin or lacosamide tablet (150 mg). At set time points the hypercapnic ventilatory response will be measured, relief of nociception, pupil diameter and several side effects other than respiratory depression such as sedation, nausea and vomiting. There will be a washout period of 7 days between study visits with the study ending after 2 visits.

Breathing tests: Breathing tests are so-called rebreathing tests in which subjects inhale 7% CO2 in oxygen from a 4-6 L rebreathing bag. By rebreathing carbon dioxide for 3-5 minutes the hypercapnic ventilatory response will be obtained. Ventilation will be measured via the pneumotachograph system.

Electrical pain test: A locally designed and manufactured transcutaneous electrical stimulation device is used to create a constant current electrical stimulus train (stimulation at 20 Hz, pulse duration 0.2 ms). The device is attached to two surface electrodes that are applied on the skin over the tibial bone of the non-dominant side. The current over the electrodes is increased from 0 mA at a rate of 0.5 mA/s, to a maximum of 128 mA. The subjects are instructed to indicate when the stimulation becomes painful (electrical pain threshold, EPTh) by pressing a button on a control box. By pressing a second button, the subjects will end the stimulus train when the pain is perceived as intolerable (electrical pain tolerance, EPTol).

Pressure pain test: a pressure pain stimulus will be applied on the skin area (1 cm2) between thumb and index finger, by using the Wagner Instruments FDN 200 Algometer. Subjects will indicate when the pressure stimulus becomes painful (pain threshold) after which the stimulus is stopped. The pressure necessary to induce pain will be recorded. The pressure pain test will follow the electrical pain test by 5-10 min.

Questionnaires: the subjects will be queried using Visual Analogue Scales from 0-10 cm (range from no effect to most severe effect), for sedation, nausea and vomiting. Additionally, the occurrences of vomiting will be counted.

Pupil diameter: At 30-min intervals, the pupil diameter will be measured using a handheld pupillometer (Neuroptics PLR-3000 pupillometer).

Amendment:

In the study, the effect of two drugs are compared, lacosamide and pregabalin, on top of 10 mg oxycodone, on the ventilatory control system. In order to get an impression of the effect of 10 mg oxycodone per se, one open label arm of just 10 mg oxycodone was added. The reason for this is many-fold:

1. It will give an indication of the effect of 10 mg oxycodone on the hypercapnic ventilatory response;
2. It will allow an indication of any difference in effect relative to oxycodone + lacosamide and oxycodone + pregabalin. Note that a formal statistical analysis between just oxycodone and oxycodone + lacosamide or oxycodone + pregabalin will not be performed. The just oxycodone data will be presented as mean ± 95% confidence interval and there will be visually determined whether the mean data from oxycodone + lacosamide and oxycodone + pregabalin fall out of the confidence interval of just oxycodone;

Since the procedures in this third arm will be identical to the two blinded arms, there will be no change to any of the procedures apart from not administering any lacosamide or pregabalin. Hence, there are no other changes to the protocol than the addition of one additional open label arm.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years,
* body mass index < 30 kg.m-2,
* able to understand the written informed consent form,
* able to communicate with the staff,
* able and willing to complete the study procedures,
* signed the informed consent form.

Exclusion Criteria:

* Presence or history of any medical or psychiatric disease (incl. a history of substance abuse, anxiety, or the presence of a painful syndrome such as fibromyalgia);
* Use of any medication in the three months prior to the study which may influence the outcome of the study as judged by the investigator;
* Use of more than 21 alcohol units per week;
* A positive urinary drug test or a breath alcohol test at screening or on the morning of the experiment;
* Pregnancy, lactating or a positive pregnancy test on the morning of the experiment;
* Participation in another drug trial in the 60 days prior to dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
Ventilation | Study day 1
  The primary endpoint of the study is the change in ventilation at an increased level of CO2
Ventilation | Study day 2
  The primary endpoint of the study is the change in ventilation at an increased level of CO2

SECONDARY OUTCOMES:
Level of sedation | Study day 1
  The subjects will be queried using Visual Analogue Scales from 0-10 cm (range from no effect to most severe effect), every hour after dosing up to 8h
Pain relief | Study day 1
  The relief of pain is measured using a painful stimulus (eg pressure pain)
Occurence of nausea/vomiting | Study day 1
  The subjects will be queried using Visual Analogue Scales from 0-10 cm (range from no effect to most severe effect).
pupil diameter | Study day 1
  Measurement of pupil diameter following drug intake.
Baseline ventilation | Study day 1
  Minute ventilation in L/min prior to increasing inhaled CO2.

CONTACTS AND LOCATIONS:
Overall Officials: Marieke Niesters, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT05598905/SAP_000.pdf